CLINICAL TRIAL: NCT05366530
Title: IdeNtification of SPecific EleCTrophenotypes in Atrial Fibrillation
Brief Title: Specific Electrophenotypes in Atrial Fibrillation
Acronym: INSPECT-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21HH7349
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarkers, electrocardiographic imaging, intracardiac electrograms, cardiac magnetic resonance imaging — ECGi is a non-invasive body surface mapping technique that collects electrocardiographic data using 252 leads, and combines it with subject specific anatomic data acquired from cross sectional imaging to recreate epicardial electrograms.

SUMMARY:
This study will investigate a common heart rhythm disturbance (arrhythmia), atrial fibrillation (AF), to improve understanding of how best to treat it in different patients. Direct current cardioversion (DCCV) is a procedure that can revert the heart to a normal rhythm, however almost all patients will only have a transient benefit, and their heart will return to the abnormal rhythm, AF. Ablation is an invasive procedure that creates scar tissue within the heart to reduce the arrhythmias, with a longer lasting effect than DCCV. It has been used with success in AF that occurs occasionally (paroxysmal) but is not as effective in AF that is more long-lasting, also known as persistent AF. Persistent AF is major cause of symptoms of breathlessness and palpitations and significantly increases the risk of stroke. Doctors are unable to accurately predict which patients will benefit most from an ablation, this can lead to as many as 50% of patients not benefitting from the procedure. The aim is to better predict which patients will benefit from an ablation. The study will include patients undergoing AF ablation or DCCV and perform additional tests including blood tests a heart MRI scan, a special type of heart tracing with up to 252 points and a short period of extra recordings from within the heart during the ablation procedure. Several techniques will be used to analyse this data, including machine learning, to develop a means predict which patients will benefit the most from the ablation procedure, without needing to use any recordings from within the heart.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for catheter mapping/ablation for arrhythmias or direct current cardioversion for atrial fibrillation
* Signed Informed Consent

Exclusion Criteria:

* Severe cerebrovascular disease
* Moderate to severe renal impairment (eGFR < 30)
* Active gastrointestinal bleeding
* Active infection or fever
* Short life expectancy
* Significant anaemia
* Severe uncontrolled systemic hypertension
* Severe electrolyte imbalance
* Congestive heart failure - NYHA Class IV
* Recent myocardial infarction
* Bleeding or clotting disorders
* Uncontrolled diabetes
* Inability to receive IV or oral Anticoagulants
* Unable to give informed consent
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing direct current cardioversion (DCCV) or catheter ablation for atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation | 1 year
  Percentage of patients who do not have a recurrence of atrial fibrillation

SECONDARY OUTCOMES:
Atrial fibrillation burden | 1 year
  Mean number of episodes of atrial fibrillation
Atrial fibrillation related symptoms and quality of life | 1 year
  Mean Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) score
Health related quality of life | 1 year
  Mean Short Form 36 (SF-36) score

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided